CLINICAL TRIAL: NCT04526405
Title: Study on the Frequency of COVID-19 Antibodies in Patients With Hereditary Hematological Diseases Subject to Chronic Transfusion Support.
Brief Title: Frequency of COVID-19 Antibodies in Patients With Hereditary Hematological Diseases
Acronym: ThalaCoV
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: ThalaCoV
Record Dates: First submitted 2020-08-06; First posted 2020-08-25 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Thalassemia Major; Covid19
MeSH Terms: conditions — beta-Thalassemia; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 S1/S2 IgG — SARS-CoV-2 S1/S2 IgG analysis

SUMMARY:
In Italy there are about 5000 patients with dependent transfusion thalassemia (source Italian Thalassemia and Hemoglobinopathies - SITE) and a smaller number, currently not definable, of patients with sickle cell anemia in chronic transfusion.

A recent study in the Lombardy region identified the positivity of anti-Covid-19 antibodies in 4.5-7% of asymptomatic donors (Valenti L et al). As already known, a preliminary study conducted in Italy (Motta I et al, Hussain FA et al, Taher A et al) reported only 11 cases of symptomatic infection all with benign evolution. Currently there are 15 reported cases (12 thalassemias and 3 sickle cell anemias). 75% of the cases have been identified in Lombardy.

Our hypothesis is that in a percentage of polytransfused patients a transmission of the virus may have developed that stimulated the production of protective antibodies. This could be an explanation of the low contagiousness and severity of the infection in polytransfused patients. Currently no data are available for this purpose.

This study will be conducted in collaboration with the Microbiology Unit and involves the determination of SARS-CoV-2 antibodies (anti-s1 and s2) by CLIA method with a high sensitivity (94.7%) and specificity (98.5%).

DETAILED DESCRIPTION:
INTRODUCTION In Italy there are about 5000 patients with dependent transfusion thalassemia (source Italian Thalassemia and Hemoglobinopathies - SITE) and a smaller number, currently not definable, of patients with sickle cell anemia in chronic transfusion.

These patients, as patients with chronic diseases, many of which also splenectomized, are generally considered to be at greater risk of infection and complications in the event of an infection.

However, preliminary studies in patients with thalassemia and sickle cell anemia do not seem to confirm these assumptions about the COVID-19 pandemic (Motta I et al, Hussain FA et al, Taher A et al). On the basis of these data, it was hypothesized that the chronic inflammatory background, the hemolytic and anemic status of these patients could have a favorable and protective influence on the risk of fatal COVID-19 infections (Roy NBA et al).

A recent study in the Milan area identified the positivity of anti-Covid-19 antibodies in 4.4-10.8% of asymptomatic donors (Valenti L et al).

TARGETS In this study, the presence of COVID-19 IgG antibodies will be assessed in all transfusion dependent patients affected by thalassemia, Blackfan-Diamond anemia, sickle cell anemia and other chronic anemias, related to the ASST-Monza Rare Disease Center, S. Gerardo and all residents in the provinces of Monza-Brianza, Como, Lecco, Varese and Milan. Of these patients, 15% experienced potentially suspect symptoms of infection, albeit mildly overall, but only 5 patients performed the nasal swab which tested positive in one case.

The study should be considered as a pilot and preliminary study since no data are available. The primary objective is to define the transfusion risk as a source of contact with the virus in patients subject to multiple transfusions (every 2-3 weeks for a total of about 300 units of blood used per month). Based on the results, further information on the exposure of these patients to COVID-19 infection may be obtained.

DESIGN This is a study with use of biological material. All patients suffering from hereditary transfusion anemias or who have undergone recurrent transfusion procedures belonging to the Rare Disease Center of ASST Monza will be enrolled in the study. The patients will be enrolled in the study when consent is obtained. A serum sample will be analyzed for anti-COVID-19 antibodies and if the result is positive, the nasal swab will be performed. If the outcome of the swab is positive, the patient must undergo quarantine and follow the national protocol. Only demographic data will be collected and only the value of antibodies to COVID-19 as biochemical data.

METHODS Serological test is based on the identification of COVID-19 antibodies (anti-s1 and -s2) by CLIA method. It has a high sensitivity (97.4%) and specificity (98.%). Although the test has a high concordance value (> 95%), it is not possible to consider if the positive subjects have neutralizing antibodies for the virus. In the case of a positive test, the molecular test for diagnostic confirmation is provided.

The analysis will be carried out at the ASST-Monza Microbiology Laboratory - S. Gerardo Hospital (Primary: Dr. Annalisa Cavallero) and an aliquot of serum will be kept at the Cytogenetics and Medical Genetics Laboratory for 1 year after the end of the study.

EXPECTED RESULTS Based on the few data available in Italy, the investigator foresees 5-10% of positive subjects.

SAMPLE SIZE AND STATISTICAL ANALYSIS All 81 transfusion dependent patients belonging to the Rare Disease Center of ASST-Monza, S. Gerardo Hospital will be included in the study and for this reason a formal calculation of sample size has not been performed.

The statistical analysis will be substantially descriptive and it will use appropriate central tendency and dispersion measures for quantitative variables, while absolute and relative frequencies will be used for qualitative variables. The estimates of the primary endpoint relating to the percentage of transfusion-dependent patients tested positive will be reported with their respective 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inherited dependent transfusion anemias (thalassemia major and intermediate, sickle cell anemia and Blackfan-Diamond anemia) or undergoing recurrent transfusion procedures (erythro-exchange in sickle cell anemia), belonging to the Rare Disease Center - ASST-Monza, Hospital S Gerardo.
* Age greater than or equal to 18 years.

Exclusion Criteria:

* No exclusion criteria are expected apart from patients' refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Transfusion dependent patients affected by thalassemia, Blackfan-Diamond anemia, sickle cell anemia and other chronic anemias, belonging to the ASST-Monza Rare Disease Center, S. Gerardo Hospital and all residents in the provinces of Monza-Brianza, Como, Lecco, Varese and Milan.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Positive subjects | 2 months
  On the basis of the few data available in Italy, the investigator foresees 5-10% of positive subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Monza - Ospedale San Gerardo, Monza, MB, Italy

REFERENCES:
- [Result] Hussain FA, Njoku FU, Saraf SL, Molokie RE, Gordeuk VR, Han J. COVID-19 infection in patients with sickle cell disease. Br J Haematol. 2020 Jun;189(5):851-852. doi: 10.1111/bjh.16734. Epub 2020 May 8. No abstract available. PMID 32314798
- [Result] Motta I, Migone De Amicis M, Pinto VM, Balocco M, Longo F, Bonetti F, Gianesin B, Graziadei G, Cappellini MD, De Franceschi L, Piga A, Forni GL. SARS-CoV-2 infection in beta thalassemia: Preliminary data from the Italian experience. Am J Hematol. 2020 Aug;95(8):E198-E199. doi: 10.1002/ajh.25840. Epub 2020 May 6. No abstract available. PMID 32311145
- [Result] Roy NBA, Telfer P, Eleftheriou P, de la Fuente J, Drasar E, Shah F, Roberts D, Atoyebi W, Trompeter S, Layton DM, Lugthart S, Stuart-Smith S, Chakravorty S, Wright J, Porter J, Inusa B, Howard J; National Haemoglobinopathy Panel. Protecting vulnerable patients with inherited anaemias from unnecessary death during the COVID-19 pandemic. Br J Haematol. 2020 May;189(4):635-639. doi: 10.1111/bjh.16687. Epub 2020 May 10. PMID 32330288
- [Result] Taher AT, Bou-Fakhredin R, Kreidieh F, Motta I, De Franceschi L, Cappellini MD. Care of patients with hemoglobin disorders during the COVID-19 pandemic: An overview of recommendations. Am J Hematol. 2020 Aug;95(8):E208-E210. doi: 10.1002/ajh.25857. Epub 2020 May 21. No abstract available. PMID 32394480
- [Result] Valenti L, Bergna A, Pelusi S, Facciotti F, Lai A, Tarkowski M, Berzuini A, Caprioli F, Santoro L, Baselli G, Della Ventura C, Erba E, Bosari S, Galli M, Zehender G, Prati D. SARS-CoV-2 seroprevalence trends in healthy blood donors during the COVID-19 Milan outbreak. medRxiv doi.org/10.1101/2020.05.11.20098442.